CLINICAL TRIAL: NCT04553653
Title: Improving Acute Hypertension Management Through Emergency Department Checklist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Aga Khan University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00195002; 5R21TW011175-02 (NIH)
Record Dates: First submitted 2020-09-11; First posted 2020-09-17 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Hypertension; Hypertensive Crisis; Hypertensive Emergency
Keywords: checklist; emergency department
MeSH Terms: conditions — Hypertension; Hypertensive Crisis; Emergencies | interventions — Checklist

STUDY DESIGN:
Intervention Model Description: This will be a before-after study. Baseline data capturing care and the outcomes of patients presenting with acute severe hypertension will be collected. A checklist will be developed and implemented and a post-implementation data collection will be conducted using the same tool as prior to the intervention.
Who Masked: Participant
Masking Description: Participants will be masked. Investigators and care providers are not masked due to the obvious design and logistics challenges.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (No Intervention): Data on diagnosis and care of patients presenting with acute severe hypertension will be collected at baseline (prior to the implementation of a checklist)
- Intervention arm (Experimental): The intervention arm will be enrolled after the checklist implementation.
  Interventions: Other: checklist

INTERVENTIONS:
Other: checklist — The checklist will be implemented and healthcare providers use the checklist to manage the patients.
  Arms: Intervention arm

SUMMARY:
The investigators hypothesize that the implementation of a checklist in acute severe hypertension would result in improving short and long-term outcomes of patients with acute severe hypertension treated in the emergency department (ED). The investigators hypothesize that in the short-term, a checklist would improve the diagnosis and management of end-organ damage as well as reduce the length of stay of acute severe hypertensive patients in the ED. The investigators hypothesize that the checklist will result in better compliance with anti-hypertensive medications than without the checklist at six-month post-discharge.

DETAILED DESCRIPTION:
Hypertension is a global public health issue and results in over 10 million deaths every year. The disease affects one-third of people living in low- and middle-income countries (LMICs) and contributes to half of all productivity losses in LMICs due to non-communicable diseases. Though hypertension often presents as a chronic asymptomatic illness, hypertension-related emergencies represent a significant burden to the health care system. Acute severe hypertension [i.e., systolic blood pressure (SBP) ≥ 180 mmHg or diastolic blood pressure (DBP) ≥ 110 mmHg] make up to 5% of all emergency admission. One-third of these patients present with end-organ damage; a condition called a hypertensive crisis. More worrisome is the fact that a number of ED visits, as a result, severe acute hypertension and hypertensive crises have almost tripled between 2006 and 2013 in the US. Treatment approaches to managing acute severe hypertension (~5% of ED patients) are largely unclear and only 6% of ED patients with acute severe hypertension receive appropriate work-up for the end-organ damage, indicating a huge care gap. One approach, which has been used successfully in managing other complex and critical conditions, is the use of checklists. Checklists are a listing of actions to be performed in a given clinical setting with the aim of improving adherence to standards, reducing errors and thus improving patient outcomes. The investigators hypothesize that the use of a Checklist, if appropriately implemented, can lead to an improvement in the care of patients presenting with hypertensive crisis. During this study, the investigators will measure the prevalence of acute severe hypertension and assess the current quality of care for these patients. This will be followed by the development of a checklist for the management of the hypertensive crises in the ED. The investigators will follow these patients to see the impact of the checklist on the quality of care and long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults who visit the Aga Khan University Hospital Emergency Department with acute severe hypertension
* able to provide consent to participate
* Age >25 years of age
* Meeting the criteria of acute severe hypertension (SBP>180 and DBP>110).

Exclusion Criteria:

* Patients not providing consent or are unconscious are excluded from participation.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1161 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in frequency of diagnosis of hypertensive emergency | Baseline and 6 months after checklist implementation
  The frequency of correct diagnosis of hypertensive emergency in patients with severe hypertension with evidence of end-organ damage in the ED before and after the implementation of the checklist.

SECONDARY OUTCOMES:
Change in the use of appropriate medications for treatment of hypertensive emergency | Baseline and 6 months after checklist implementation
  We will measure the compliance with the hypertensive emergency treatment protocol before and after implementation of the checklist.

OTHER OUTCOMES:
Compliance with chronic treatment of hypertension as assessed through a phone call | Up to 6 months post discharge from the emergency department
  We will follow up our patients on phone to assess their compliance with the use of antihypertensive medications.

CONTACTS AND LOCATIONS:
Overall Officials: Junaid A Razzak, Principal Investigator — Johns Hopkins University
Locations (1):
- Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No